CLINICAL TRIAL: NCT04838652
Title: Phase II Trial of Pembrolizumab in Combination With Salvage Chemotherapy for First-relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Pembrolizumab in Combination With Salvage Chemotherapy for First-relapsed or Refractory Classical Hodgkin Lymphoma
Acronym: Pembro-CORE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-3942
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — pembrolizumab; Drug Therapy; Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus Chemotherapy (Experimental): All patients will receive 1 dose of 200 mg pembrolizumab IV as single agent upfront, followed by 2 cycles of IV P-ICE (pembrolizumab, ifosfamide, carboplatin, etoposide) and a PET/CT-based restaging. Following a PET-guided treatment strategy, patients will then receive either another 2 cycles of IV P-ICE in case of a negative PET (i.e., Deauville score 1-3), or 2 to 4 cycles of IV P-DHAP (pembrolizumab, dexamethasone, cytarabine, cisplatin) in case of a positive PET (i.e., Deauville score > 3). After completion of treatment with P-ICE or P-DHAP, respectively, patients will receive a consolidation therapy with pembrolizumab for another 6 cycles. In case of non-CR after at least 4 cycles of combination therapy (4x P-ICE or 2x P-ICE + 2x P-DHAP), physicians may decide to go for HDCT or an alternative standard of care treatment option.
  Interventions: Drug: Pembrolizumab plus Chemotherapy (ICE or DHAP)

INTERVENTIONS:
Drug: Pembrolizumab plus Chemotherapy (ICE or DHAP) — Pembrolizumab (200mg) alone or in combination with ICE (or DHAP in case of PET positive findings after P-ICE) will be admistered. 6 additional courses of pembrolizumab will be administered after the completion P-ICE or P-DHAP

SUMMARY:
The aim of this trial is to develop an effective and well-tolerated regimen for treatment of r/r cHL by introducing the anti-PD-1 antibody pembrolizumab and adding it to well-established chemotherapy regimens (ICE, DHAP). Synergistic effects of conventional agents with checkpoint inhibition may facilitate a highly effective therapy with limited toxicity, which might eventually substitute the very toxic high-dose chemotherapy (HDCT).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed first relapse of cHL or primary refractory cHL

Exclusion Criteria:

* Nodular lymphocyte-predominant Hodgkin lymphoma or composite lymphoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Complete Metabolic Response Rate (CMR) | after completion of P+chemotherapy, an average of 3 months
  The proportion of patients with a Deauville score of 1-3 in the centrally reviewed restaging after treatment with 1 x pembrolizumab + 4 cycles of pembrolizumab and chemotherapy combined (4x P-ICE or 2x P-ICE + 2x P-DHAP)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — 1st Department of Medicine, Cologne Universit Hospital
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany